CLINICAL TRIAL: NCT06085222
Title: Refinement and Testing of a Brief Computerized and Smart Phone-based Intervention for Stress in Regular Cannabis Users
Brief Title: Evaluation of a Brief Computerized and Smart Phone-based Intervention for Stress in Regular Cannabis Users
Acronym: DISC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Northwestern University (Other); Duke University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Rick James Macatee, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00006346; 1R34DA057733-01A1 (NIH)
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cannabis Use Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Engagement Distress Tolerance Intervention (Experimental): The experimental intervention (single 2.5 hour session) is comprised of video-delivered psychoeducation, adaptive skill practice, and emotional exposure. During exposure, a sequence of percussive sounds accompanied by a visual depiction of the participant's skin conductance level during exposure will be presented at the moment the participant's skin conductance returns to the relaxation baseline value. These images/sound will be intermittently sent to the participant's smart phone during the smart phone portion of the intervention.
  Interventions: Behavioral: Emotional Engagement Distress Tolerance Intervention
- Health Education Intervention (Placebo Comparator): The health education control intervention is a single 2.5 hour computerized session. It is comprised of audio-narrated videos on healthy habits and self-care in the domains of sleep, nutrition, hygiene, and physical exercise. The same sequence of percussive sounds used in the Emotional Engagement Distress Tolerance Intervention is presented alongside summary slides presenting key points on healthy habits and self-care. These images/sound will be intermittently sent to the participant's smart phone during the smart phone portion of the intervention.
  Interventions: Behavioral: Health Education Intervention

INTERVENTIONS:
Behavioral: Emotional Engagement Distress Tolerance Intervention — 2.5 hour computerized intervention with smart phone support focused on building tolerance of emotional distress
  Arms: Emotional Engagement Distress Tolerance Intervention
Behavioral: Health Education Intervention — 2.5 hour computerized intervention with smart phone support focused on building healthy habits that support stress management
  Arms: Health Education Intervention

SUMMARY:
The prevalence of daily cannabis use and Cannabis Use Disorder (CUD) has increased in the United States over the past two decades. Brief, computerized harm reduction interventions that target specific high-risk CUD populations could be an efficient approach to reducing CUD. Distress intolerance , which refers to the tendency to negatively appraise and escape aversive emotional states, is a risk factor associated with stress-related cannabis use motivation and CUD severity/chronicity. Thus, a brief, accessible, low-cost intervention that reduces distress intolerance in those with CUD and elevated distress intolerance could have a significant public health impact. This proposed project aims to optimize an existing two-session computerized distress tolerance intervention and test its impact on distress intolerance and cannabis use outcomes in a randomized controlled trial. Specifically, the intervention will be condensed to one-session, its active ingredient bolstered, and augmented with smart phone-delivered therapy reminders. After obtaining feedback on the modified Emotional Engagement Distress Tolerance Intervention in a small sample, the intervention's efficacy compared to a stringent, credible, time-matched health education control intervention will be tested in a randomized controlled trial in 80 cannabis users with CUD and high distress intolerance. Distress intolerance, cannabis use, and psychosocial functioning outcomes will be evaluated. As an exploratory aim, a wristworn device will be used to measure objective stress responding in the real-world during the intervention period. Our central hypothesis is that, compared to a control intervention, the Emotional Engagement Distress Tolerance Intervention will produce superior reductions distress intolerance, stress-related cannabis use motivation, disordered cannabis use, and psychosocial functioning.

DETAILED DESCRIPTION:
The prevalence of daily cannabis use and Cannabis Use Disorder (CUD) has increased in the United States over the past two decades. Brief, computerized harm reduction interventions that target specific high-risk CUD populations could be an efficient approach to reducing CUD. Distress intolerance, which refers to the tendency to negatively appraise and escape aversive emotional states, is a risk factor associated with stress-related cannabis use motivation and CUD severity/chronicity. Thus, a brief, accessible, low-cost intervention that reduces distress intolerance in those with CUD and elevated distress intolerance could have a significant public health impact. This proposed Stage I project aims to modify an existing two-session computerized distress tolerance intervention to optimize emotion regulation learning/generalization and test its impact on distress intolerance and cannabis use outcomes in a randomized controlled trial. Specifically, the intervention will be condensed to one-session and its imaginal exposure module will be modified to shape emotional engagement with the aim of maximizing within-session habituation, which will be signaled with a novel audio/visual cue (habituation cue). Habituation cues will then be delivered in just-in-time text message reminders triggered by naturalistic distress reported via ecological momentary assessment. After obtaining feedback on the modified Emotional Engagement Distress Tolerance Intervention in a small sample, the intervention's efficacy compared to a stringent, credible, time-matched health education control intervention will be tested in a randomized controlled trial in 80 cannabis users with CUD and high distress intolerance. To measure the intervention's mechanistic target engagement, multi-method distress intolerance assessments will be administered through four-month follow-up. To measure the intervention's impact on cannabis use, stress-related cannabis use motivation (lab stress- elicited craving and neurophysiological drug cue reactivity, ecological momentary assessment of stress-elicited cannabis use) will be assessed through the intervention period. Interviewer-assessed cannabis use frequency, CUD severity, and urinary THC metabolite concentration will be measured through 4-month follow-up. Quality of life and anxiety/depression symptoms will also be measured as secondary outcomes through 4-month follow-up. As an exploratory aim, a wristworn device will be used to measure ambulatory physiology during a portion of the intervention period to evaluate the feasibility of detecting heightened real- world distress based on objective indicators. Our central hypothesis is that, compared to a control intervention, the Emotional Engagement Distress Tolerance Intervention will produce superior reductions in multi-method assessments of distress intolerance, stress-related cannabis use motivation, disordered cannabis use, and psychosocial functioning. Successful completion of the proposed aims will (1) justify a subsequent Stage II trial, and (2) inform efforts to integrate the just-in-time habituation reminders with wearable technology in order to increase emotion regulation generalization opportunities and decrease participant report burden.

ELIGIBILITY:
Inclusion Criteria:

* Cannabis is the primary substance of abuse.
* Clinical-level Distress intolerance Index score.
* Current Cannabis Use Disorder diagnosis.
* Near-daily to daily cannabis use in past-month and past 3 months.
* Positive urine screen for THC
* Detectable skin conductance level
* Owns a smart phone
* Primary smoked/vaporized delta-9 or delta-8 THC user

Exclusion Criteria:

* Presence of acute/major psychiatric disturbance
* Current pregnancy
* Change in psychotropic medication within the past month
* Concurrently receiving treatment for cannabis use
* Concurrently receiving dialectical behavior therapy or exposure-based therapy for emotional disorders
* Planning to immediately quit using cannabis
* EEG contraindications
* Kidney disease

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Therapy Evaluation Questionnaire | Immediately after intervention session
  acceptability/feasibility (credibility subscale range 3-27; expectancy item range 0%-100%; higher scores indicate better outcome)
Treatment Satisfaction Questionnaire | Post-Intervention (20 days after intervention session)
  acceptability/feasibility (range 0-84; higher scores indicate better outcome)
Change in perceived distress intolerance from baseline through follow-up | Baseline, Mid-Intervention (10 days after intervention session), Post-Intervention (20 days after intervention session), One-Month Follow-up, Four-Month Follow-up
  Distress Intolerance Index (range 0-40; higher scores indicate worse outcome) to assess perceived distress intolerance via self-report
Change in behavioral distress intolerance from baseline through follow-up | Baseline, Mid-Intervention (10 days after intervention session), Post-Intervention (20 days after intervention session), One-Month Follow-up, Four-Month Follow-up
  Mirror-Tracing Persistence Task to assess behavioral distress intolerance via computerized task
Change in laboratory stress-induced cannabis craving from baseline through post-intervention | Baseline, Post-Intervention (20 days after intervention session)
  Change in Marijuana Craving Questionnaire (range 11-77; higher scores indicate worse outcome) after Mannheim Multicomponent Stress Test at post-intervention compared to baseline
Change in laboratory stress-induced neural reactivity to cannabis cues (assessed via the electroencephalography [EEG]-recorded late positive potential) from baseline through post-intervention | Baseline, Post-Intervention (20 days after intervention session)
  Change in Late Positive Potential to Cannabis Cues after Mannheim Multicomponent Stress Test at post-intervention compared to baseline
Change in real-world stress-elicited cannabis use from baseline to post-intervention | Baseline, Mid-Intervention (10 days after intervention session), Post-Intervention (20 days after intervention session)
  Change in stress->cannabis use slopes derived from ecological momentary assessment from baseline through post-intervention
Change in cannabis use frequency from baseline through follow-up | Baseline, Post-Intervention (20 days after intervention session), One-Month Follow-up, Four-Month Follow-up
  Change in cannabis use frequency (measured via timeline follow-back) from baseline through four-month follow-up
Change in urine tetrahydrocannabinol [THC] metabolite concentration from baseline through follow-up | Baseline, Mid-Intervention (10 days after intervention session), Post-Intervention (20 days after intervention session), One-Month Follow-up, Four-Month Follow-up
  Change in urinary THC metabolite concentration (measured via ultra high performance liquid chromatography [UHPLC]) from baseline through four-month follow-up
Change in self-reported cannabis use problems from baseline through follow-up | Baseline, Post-Intervention (20 days after intervention session), One-Month Follow-up, Four-Month Follow-up
  Change in Marijuana Problems Scale (range 0-38; higher scores indicate worse outcome) from baseline through follow-up
Change in Cannabis Use Disorder symptoms from baseline through follow-up | Baseline, Four-Month Follow-up
  Change in interviewer-assessed Cannabis Use Disorder criteria (range 0-11; higher scores indicate worse outcome) from baseline to four-month follow-up
Change in Cannabis Demand from baseline to post-intervention | Baseline, Post-Intervention (20 days after intervention session)
  Change in Omax, Breakpoint, and Elasticity derived from Marijuana Purchase Task (higher OMax/Breakpoint and lower Elasticity indicate worse outcome) at post-intervention compared to baseline
Change in cannabis use quantity from baseline to post-intervention | Baseline, Post-Intervention (20 days after intervention session), One-Month Follow-up, Four-Month Follow-up
  Change in cannabis use quantity (measured via timeline follow-back) from baseline through four-month follow-up

SECONDARY OUTCOMES:
Change in quality of life from baseline through follow-up | Baseline, Post-Intervention (20 days after intervention session), One-Month Follow-up, Four-Month Follow-up
  Change in self-reported quality of life (measured via Quality of Life Enjoyment and Satisfaction Questionnaire Short-Form; range 16-80; lower scores indicate worse outcome) from baseline through follow-up
Change in depression and anxiety from baseline through follow-up | Baseline, Post-Intervention (20 days after intervention session), One-Month Follow-up, Four-Month Follow-up
  Change in self-reported depression and anxiety (measured via Hospital Anxiety and Depression Scale [range 0-21 for each subscale; higher scores indicate worse outcomes) from baseline through follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Macatee, PhD, Principal Investigator — Florida State University
Locations (1):
- The BRAINS Lab at Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No